CLINICAL TRIAL: NCT01100060
Title: A Phase 1, Open-Label, Randomized, Single Dose, Parallel Design Study To Estimate The Relative Bioavailability Of Co Administered Formulations Of Azithromycin Microsphere (AZ) And Chloroquine Test Formulation (CQ) Compared With Co Administered Immediate Release Individual AZ And CQ Tablets In Healthy Adult Subjects
Brief Title: A Phase 1 Study To Estimate The Relative Bioavailability Of Co-Administered Formulations Of Azithromycin Microsphere And Chloroquine Test Formulation Compared With Co-Administered Immediate Release Individual Azithromycin And Chloroquine Tablets In Healthy Adult Subjects
Acronym: AZCQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A0661195
Record Dates: First submitted 2010-03-26; First posted 2010-04-08 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Malaria Prophylaxis
Keywords: Azithromycin; chloroquine; microsphere; pharmacokinetics; bioavailability
MeSH Terms: interventions — Azithromycin; Microspheres; Dosage Forms; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Co-administer the test chloroquine (CQ) formulation (620 mg CQ base) plus microsphere azithromycin (AZ) (2000 mg) on Day 1.
  Interventions: Drug: azithromycin (AZ) microsphere; Drug: test chloroquine (CQ) formulation
- Group 2 (Active Comparator): Co-administer the individual tablets of CQ 2 x 500 mg (600 mg CQ base) tablets plus AZ IR 4 x 500 mg tablets on Day 1.
  Interventions: Drug: azithromycin (AZ); Drug: chloroquine (CQ)

INTERVENTIONS:
Drug: azithromycin (AZ) microsphere — AZ microsphere (2000 mg) single dose on Day 1.
  Other Names: Zmax
  Arms: Group 1
Drug: test chloroquine (CQ) formulation — Test CQ formulation, 620 mg CQ base, single dose on Day 1.
  Arms: Group 1
Drug: azithromycin (AZ) — AZ IR 4 x 500 mg tablets, single dose on Day 1.
  Other Names: Zithromax
  Arms: Group 2
Drug: chloroquine (CQ) — CQ 2 x 500 mg (600 mg CQ base) tablets, single dose on Day 1
  Other Names: Aralen
  Arms: Group 2

SUMMARY:
Estimate the relative bioavailability of co-administered azithromycin microsphere (2000 mg) and the chloroquine (620 mg CQ base) test formulation compared to co-administered immediate release individual tablets of azithromycin (2000 mg) and chloroquine (600 mg CQ base) in healthy adult subjects.

DETAILED DESCRIPTION:
Evaluate the relative bioavailability, assessment of the safety and tolerability of azithromycin microsphere and the chloroquine test formulation compared to immediate release individual tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of febrile illness within 5 days prior to first dose.
* Treatment with azithromycin within the past 30 days or with chloroquine within the past 45 days.
* Known immediate family history of prolonged QT Syndrome, serious ventricular arrhythmia, or sudden cardiac death. "Immediate" is considered "first degree".
* Known allergy to macrolide antibiotics (eg, erythromycin, clarithromycin, azithromycin) or chloroquine (or other 4 aminoquinolines) or severe allergic reaction to any drug in the past (eg, difficulty breathing, anaphylaxis).
* History of intolerance to azithromycin or chloroquine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
AUClast of azithromycin and chloroquine | Through Day 5

SECONDARY OUTCOMES:
Tmax and Cmax of azithromycin and chloroquine. | Through Day 5
AUClast, Tmax, and Cmax of desethylchloroquine. | Through Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661195&StudyName=A%20Phase%201%20Study%20To%20Estimate%20The%20Relative%20Bioavailability%20Of%20Co-Administered%20Formulations%20Of%20Azithromycin%20Microsphere%20And%20Chloroquine%20Test%20